CLINICAL TRIAL: NCT02882360
Title: The Use of Antimicrobial Gauze in Pregnant Women Undergoing C-section With BMI >40 to Decrease Wound Complications by 6 Weeks postpartum--a Small Feasibility Study
Brief Title: Kerlix for Pregnant Women With Elevated BMI to Prevent Wound Infection by 6 Weeks Post Partum
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Debbie Penava, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 106708
Record Dates: First submitted 2016-05-12; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Wound Infection; Pregnancy
MeSH Terms: conditions — Obesity; Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Elective LSCS--Kerlix AMD (Experimental): Kerlix-AMD applied to wound site pre-operatively (3 days) and post-operatively for 2 weeks
  Interventions: Device: Kerlix-AMD
- Elective LSCS--Placebo (Placebo Comparator): Normal gauze applied to wound site pre-operatively for 3 days and post-operatively for 2 weeks
  Interventions: Other: placebo--normal gauze
- Labouring LSCS--Kerlix AMD (Experimental): Kerlix-AMD applied to wound post-operatively for 2 weeks
  Interventions: Device: Kerlix-AMD
- Labouring LSCS--Placebo (Placebo Comparator): Normal gauze applied to wound post-operatively for 2 weeks
  Interventions: Other: placebo--normal gauze

INTERVENTIONS:
Device: Kerlix-AMD — Application of PHMB impregnated gauze pre-operatively (for booked C-sections) and post-operatively for all patients with LSCS. Gauze to be changed daily or more frequently if damp/blood-tinged
  Arms: Elective LSCS--Kerlix AMD; Labouring LSCS--Kerlix AMD
Other: placebo--normal gauze — Application of gauze pre-operatively (for booked C-sections) and post-operatively for all patients with LSCS. Gauze to be changed daily or more frequently if damp/blood-tinged
  Arms: Elective LSCS--Placebo; Labouring LSCS--Placebo

SUMMARY:
Pregnant women with BMI>40 will be approached for participation in a study to reduce the rate of post-operative wound infection from C-section. Women will be randomized to a commonly used wound product (Kerlix-AMD) which consists of a PHMB-impregnated gauze versus normal gauze, and rates of post-operative surgical site infection will be assessed. Women with a planned procedure will also be randomized to applying Kerlix versus gauze for 3 days pre-operatively to determine if this improves outcomes as well.

DETAILED DESCRIPTION:
This study be a randomized double-blinded feasibility study to improve the rates of wound complications post-C/S in women with a BMI >40. It will be conducted out of a single tertiary care centre in London, Ontario. The women will be randomized to one of two treatment groups, either Kerlix AMD gauze or Kerlix plain gauze (Kendall, Covidien AG, Mansfield MA). This randomization will be performed by validated computer based randomization software (www.sealedenvelope.com). The patients, staff and physicians will be blinded to the assigned groups. After consenting to the study, at the time of their C/S, participants will be assigned a sealed envelope which will contain their assigned group. All patients with a BMI >40 who qualify for the study that are seen in the outpatient clinics at our centre will be approached about their participation in the study. Patients that meet the study criteria who are seen for the first time after being admitted to the labor and delivery ward will be consented for the study, and if they do not require a C/S, then this consent will be disregarded. Participants who have a planned C/S will also be randomized to receive treatment with either AMD or plain gauze for three days prior to their C/S. This requires placement of a piece of gauze, randomly assigned, under the pannus in the area of the anticipated incision. This gauze is to be changed daily for three days prior to the booked C/S. These patients will continue to receive the same gauze they were assigned to post-operatively. As part of routine care peri-operatively, all patients receive 3g of Ancef 15-60 min prior to skin incision (Ayres-de-Campos), and their skin is prepped with 2% chlorohexidine (Lee I) (2%, Laboratoire Atlas Inc, Montreal, QC) . The subcutaneous layer will be closed at the end of the case using absorbable sutures (Chelmow). The skin will be closed with a running absorbable suture in the subcuticular layer (Clay). At the end of the C/S, all patients will have their respective gauze placed over their incision, with a Tegaderm (3M Healthcare, St. Paul, MN) or pressure dressing placed on top. This outer occlusive dressing will be removed poat-operative day )POD) 1, unless it becomes saturated before then. Their gauze will be replaced daily, or more frequently if it becomes saturated. The incisions will be inspected daily by a physician while they are in hospital. The Centers for Disease Control and Prevention (CDC) Nosocomial Infections Surveillance (NNIS) system criteria will be used to diagnose wound infections. They will be discharged home with enough gauze for daily dressing changes for two weeks, as well as an information sheet outlining signs and symptoms to be aware of, or reasons to return to hospital. Their incision will be inspected by a physician at one, two and six weeks post-operatively. If at any point over the duration of the study they develop signs or symptoms of infection or any other complications, they will be investigated and treated accordingly. This may involve taking a picture of the wound to track whether or not cellulitis or infection is spreading or tracking; this will always be with your explicit consent and to track wound progression. At six weeks they will also complete a qualitative survey investigating their subjective experience with the gauze and the protocol. A cost analysis will also be performed. All data will be collected using data collection sheets. The newest version of Statistical Package for Social Sciences (SPSS) Statistical analysis software will be used to conduct data analysis, using formulas such as student t-test for continuous data and chi-squared for nominal data.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at LHSC with BMI >40

Exclusion Criteria:

* pregnant women who cannot understand English, who have a fetal demise or who have a pre-existent infected skin infection at the site of c-section

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
surgical site infection | 6 weeks
  All patients will have their wounds assessed by 6 weeks post partum to evaluate for the presence (or absence) of surgical site infection, using the Centers for Disease Control and Prevention (CDC) Nosocomial Infections Surveillance (NNIS) system criteria.

SECONDARY OUTCOMES:
patient satisfaction | 6 weeks
  patients will be surveyed on adherence and acceptability of application of gauze post c-section

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Penava, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's

IPD SHARING:
Plan to Share IPD: No